CLINICAL TRIAL: NCT00480870
Title: The Effect of Anticholinesterase Drugs on Sleep in Alzheimer's Disease Patients
Acronym: ACHALZSLEEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Walter Andre dos Santos Moraes/ MD PhD, AFIP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP nº051/99
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer Disease; Sleep Apnea, Obstructive
Keywords: Alzheimer; polysomnography; REM sleep; donepezil; sleep apnea; oxygen saturation
MeSH Terms: conditions — Alzheimer Disease; Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Donepezil

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Donepezil treated Alzheimer patients
  Interventions: Drug: donepezil
- B (Placebo Comparator): Placebo treated Alzheimer patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: donepezil — donepezil 5 mg 1 p / day for 1 month and 2p / day for 5 months on.
  Arms: A
Drug: Placebo — Placebo 1p / day for 1 month and 2 / day for 5 months on
  Arms: B

SUMMARY:
The purpose of this study is to determine the effects of the anticholinesterase drug donepezil on sleep in Alzheimer disease patients. Sleep structure and respiratory parameters will be analyzed by polysomnography.

DETAILED DESCRIPTION:
Central acting cholinesterase inhibitors are the first primary pharmacological treatment approved for Alzheimer disease, of which donepezil is the most frequently used. Multicenter studies have found little toxicity, and its side effects (diarrhea, nausea, vomiting, nightmares, among others) are mild and transient. According to the literature, cholinergic active drugs may be expected to affect REM (rapid eye movement) sleep. Another possible effect is related to respiratory parameters in patients with Alzheimer disease and obstructive sleep apnea. In fact, cholinergic activity influences the upper airway opening via central and peripheral mechanisms.

Intervention: Patients will be administered donepezil or placebo. The study has a randomized, double-blind placebo-controlled design. Complete polysomnography with REM sleep EEG spectral analysis and ADAS-cog scoring will be performed at baseline and after 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease based on the probability criteria of the Alzheimer's Disease and Related Disorders Association
* Rated 1 and 2 (mild to moderate level) on the Brazilian version of the Clinical Dementia Rating

Exclusion Criteria:

* Other causes of dementia
* Other severe medical or psychiatric disease
* Clinical indication of psychoactive drugs other than experimental drug

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 1999-04; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Polysomnography parameters: sleep structure, respiratory, limb movements | onset, 3 and 6 months of treatment

SECONDARY OUTCOMES:
Brain magnetic resonance imaging | onset
laboratory tests: hematological evaluation, creatinine, vitamin B12-folic acid, thyroid hormones, GOT, GPT, GGT, bilirubin, fasting glycemia, venereal disease research test and urine sediment | onset
electroencephalogram | onset
Mini-mental state examination | onset
IDATE | onset
Frequency bands of scalp EEG areas: overall (average of all electrodes), frontal (F3, F4, F7, F8, Fz), temporal (T3, T4, T5, T6), parietal (P3, P4, Pz), central (C3, C4, Cz), and occipital (O1, O2, Oz). | onset, 3 and 6 months of treatment
ADAS-cog scores | onset, 3 and 6 months of treatment
Clinical Dementia Rating | onset
EEG slowing ratio | onset, 3 and 6 monthes of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Walter AS Moraes, MD PhD, Principal Investigator — Associação Fundo de Incentivo a Psicofarmacologia - AFIP
Locations (1):
- Instituto do Sono, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rosa A, Poyares D, Moraes W, Cintra F. Methodology in clinical sleep research. Cell Mol Life Sci. 2007 May;64(10):1244-53. doi: 10.1007/s00018-007-6535-y. PMID 17364137
- [Background] Lucchesi LM, Pradella-Hallinan M, Lucchesi M, Moraes WA. [Sleep in psychiatric disorders]. Braz J Psychiatry. 2005 May;27 Suppl 1:27-32. doi: 10.1590/s1516-44462005000500006. Epub 2005 Jul 28. Portuguese. PMID 16082452
- [Result] Moraes Wdos S, Poyares DR, Guilleminault C, Ramos LR, Bertolucci PH, Tufik S. The effect of donepezil on sleep and REM sleep EEG in patients with Alzheimer disease: a double-blind placebo-controlled study. Sleep. 2006 Feb;29(2):199-205. doi: 10.1093/sleep/29.2.199. PMID 16494088
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083
- [Derived] Moraes W, Poyares D, Sukys-Claudino L, Guilleminault C, Tufik S. Donepezil improves obstructive sleep apnea in Alzheimer disease: a double-blind, placebo-controlled study. Chest. 2008 Mar;133(3):677-83. doi: 10.1378/chest.07-1446. Epub 2008 Jan 15. PMID 18198262